CLINICAL TRIAL: NCT07255443
Title: Intestinal Colonization With Carbapenem Resistant Enterobacteriaceae Among ICU Patients at Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Israa Ahmed abdelhalim (Other)
Responsible Party: Sponsor-Investigator, Israa Ahmed abdelhalim, Resistant doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Assiut_icu_catbapenem_2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Rate of Carbapenemase Intestinal Carrier Inside ICU
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Prospective cohort study conducted in the Adult ICU at Assiut University Hospital
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
significant benefits by providing data to improve infection control, guide early detection, and reduce CRE transmission in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)_

  * Expected ICU stay ≥48 hours -

Exclusion Criteria:

* .ICU stay <48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible adult patients admitted during the study period
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
rate of intestinal colonization with CRE | One year